CLINICAL TRIAL: NCT03517813
Title: Comparative Performance of Contrast-enhanced Spectral Mammography (CESM) and Abbreviated Breast MRI (ABMR) With Standard Breast MRI for Breast Cancer Screening
Brief Title: CESM ABMR Breast Cancer Screening Trial
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 9745; RG3016008 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2021-12488 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-03-27; First posted 2018-05-07 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer Screening

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Cohort 1: Asymptomatic women at increased risk of breast cancer referred clinically for high risk screening breast MRI or women with newly diagnosed primary unilateral breast cancer referred for evaluation of extent of disease (EOD) in the index breast and screening of the contralateral breast.
  All women enrolled on study will complete a clinical breast MRI and research contrast enhanced mammogram. Abbreviated MRI images will be extracted from the standard breast MRI exam.
  Interventions: Device: Contrast-enhanced Spectral Mammography (CESM)
- Cohort 2: Women receiving MRI for any indication and for whom percutaneous biopsy with ultrasound or MRI guidance has been recommended.
  All women enrolled on study will complete a standard breast MRI and research contrast enhanced mammogram. Abbreviated MRI images will be extracted from the standard breast MRI exam.
  Interventions: Device: Contrast-enhanced Spectral Mammography (CESM)

INTERVENTIONS:
Device: Contrast-enhanced Spectral Mammography (CESM) — Dual energy mammography images obtained after the administration of an intravenous contrast agent

SUMMARY:
This is a single institution, prospective screening trial of women at high risk for developing breast cancer, enriched with women with suspicious lesions on breast MRI which have been recommended for biopsy.

Primary Aim: Measure and compare the diagnostic performance of CESM, ABMR, and standard breast MRI, using the following performance measures: cancer detection rate (CDR), biopsy rate, and cancer yield of biopsy (also known as positive predictive value 3 or PPV3).

Secondary Aims:

1. Compare screening performance outcome measures of sensitivity, specificity, and area under the receiver operating characteristic curve (AUC) for CESM, ABMR, and standard breast MRI. This will determine the feasibility of each modality as an alternative to standard breast MRI and provide valuable pilot data for designing a larger clinical trial to evaluate non-inferiority of either or both modalities.
2. Breast cancer characteristics (size, histologic subtype, node-positivity, AJCC stage) will be assessed in the overall cohort, and stratified by mode of detection for each modality(screen-detected versus interval).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide signed declaration of informed consent or have a legally authorized representative provide signed declaration of informed consent for participation in all study procedures;
* Women aged ≥18 years at the time of enrollment
* Referred clinically for breast MRI for any indication

Exclusion Criteria:

* Known allergy or contraindication to iodinated contrast
* Are currently pregnant based on urine pregnancy test
* Have breast implants
* Are lactating

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women referred for a clinical breast MRI.
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Abnormal interpretation rate | 2 years
  Abnormal interpretation rates for each modality (CESM, abbreviated breast MRI, standard breast MRI)

SECONDARY OUTCOMES:
Biopsy rate | 2 years
  Biopsy rate will be assessed for each modality (CESM, abbreviated breast MRI, standard breast MRI)
Positive predictive value for biopsy recommendation (PPV2) | 3 years
  Positive predictive value for biopsy recommendation (PPV2) will be assessed for each modality (CESM, abbreviated breast MRI, standard breast MRI)
Negative predictive value | 3 years
  Negative predictive value will be assessed for each modality (CESM, abbreviated breast MRI, standard breast MRI)
Cancer detection rate | 3 years
  Cancer detection rate will be assessed for each modality (CESM, abbreviated breast MRI, standard breast MRI)
Sensitivity | 2 years
  Sensitivity will be assessed for each modality (CESM, abbreviated breast MRI, standard breast MRI)
Specificity | 2 years
  Specificity will be assessed for each modality (CESM, abbreviated breast MRI, standard breast MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Janie M Lee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Seattle Cancer Care Alliance, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No